CLINICAL TRIAL: NCT04043247
Title: Transcutaneous Electrical Acupoint Stimulation for Prevention of Postoperative Nausea and Vomiting: a Multicenter, Evaluator-Blind, Randomized and Controlled Study
Brief Title: Transcutaneous Electrical Acupoint Stimulation for Prevention of Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XJTU1AF2019LSK-084
Record Dates: First submitted 2019-07-29; First posted 2019-08-02 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting;TEAS
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): Same as TEAS group but without electrical stimulation
  Interventions: Device: TEAS without electrical stimulation
- TEAS Group (Experimental): Bilateral Neiguan and Zusanli acupuncture points, 2/10Hz Dense wave , 6-9mA,30min
  Interventions: Device: TEAS

INTERVENTIONS:
Device: TEAS — Bilateral Neiguan and Zusanli acupuncture points, 2/10Hz Dense wave , 6-9mA,30min
  Arms: TEAS Group
Device: TEAS without electrical stimulation — Bilateral Neiguan and Zusanli acupuncture points, with no electrical stimulation
  Arms: Control Group

SUMMARY:
Postoperative nausea and vomiting(PONV) refers to at least one nausea, retching or vomiting after operation, or any combination of the above symptoms. The incidence of PONV in high-risk patients can reach 61%-79%. PONV can not only cause dizziness and headache, but also cause disturbance of acid-base balance of water and electrolyte, wound dehiscence, formation of incisional hernia, aspiration, and aspiration pneumonia, leading to prolonged hospitalization, increased medical expenses, and reduced surgical satisfaction. At present, the guidelines for prevention and treatment of PONV and the consensus of experts suggest that identifying high-risk patients according to Apfel risk score ≥3 points, reducing baseline PONV risks, and implementing multimodal PONV prophylaxis. However, the incidence of PONV in high-risk patients is still as high as 20% even if 2-3 drugs are combined used for prevention and treatment. It is difficult to further reduce the incidence of PONV by adding different kinds or dosages of drugs, while drug-related side effects are increasing gradually. Acupuncture (electroacupuncture, transcutaneous electrical acupoint stimulationTEAS, transcutaneous electrical nerve stimulation, etc.) is a safe, effective, non-toxic side-effect non-drug treatment method. A large number of studies have confirmed that acupuncture can reduce the incidence of PONV, and it is expected to become an important supplement to drug treatment of PONV, but there are quality defects such as small sample size, inaccurate intervention and so on. At the same time, most acupuncture studies aim to compare the efficacy of PONV with drug therapy, without considering the clinical situation, using acupuncture treatment based on drug standard treatment to further reduce the incidence of PONV, thus limiting the clinical application value of acupuncture. On the basis of standardized drug prevention and treatment of PONV, TEAS will be used to further reduce the incidence of PONV and promote rapid recovery of patients. This study will strongly demonstrate that acupuncture can break through the bottleneck of drug treatment and provide evidence for the application of acupuncture in modern perioperative clinical medicine.

DETAILED DESCRIPTION:
This study intends to carry out a high-quality clinical research with design specifications, large sample, multi-center, evaluator blinded, randomized and controlled methods. From September 1, 2019 to October 30, 2020, patients undergoing laparoscopic non-gastrointestinal surgery under general anesthesia will be recruited, based on the combination of dexamethasone and 5-HT3 antagonist, the efficacy of TEAS stimulation Neiguan (P6) and Zusanli (ST36) in the prevention and treatment of PONV will be verified. In TEAS group, bilateral P6 and ST36 TEAS intervention after removal tracheal intubation and on the first day after surgery, a total of 2 times, 30 minutes each time, 2/10 Hz low frequency sparse wave, 6-9 mA. The patients will be given maximum intensity stimulation at all points during the intervention.To ensure the blindness of the evaluator, the time of evaluation will be on the afternoon of the first and the second day, and the 30 days after the operation, and three evaluations will be made. The main indicators are the incidence of PONV 24 hours after operation, and the secondary indicators are the quantitative indicators of PONV and the indicators of rapid recovery after operation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years old, BMI 15~40kg/m2, ASAI-III;
* Laparoscopic non-gastrointestinal surgery under general anesthesia;
* Postoperative Nausea and Vomiting Apfel ≥3;
* Understand and sign an informed consent form and cooperate with the intervention and evaluation;

Exclusion Criteria:

* Pregnancy, lactation period;
* Taboos of transcutaneous electrical stimulation: skin allergy, damage, infection and itching at test acupoints; allergy to tape; pacemaker implanter;
* Identify/discriminate a history of alcohol, opioids or other drugs abuse;
* Admission to ICU after surgery;
* Participation in other clinical studies within 3 months before admission to this study;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1655 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV within 24 hours | 24 hours after surgery
  Whether or not nausea or vomiting happens

SECONDARY OUTCOMES:
The first nausea | 24 hours after surgery
  the time point of the first nausea.
The first nausea's Visual Analogue Scale | 24 hours after surgery
  the Visual Analogue Scale of the first nausea : the Visual Analog Scale (VAS) is a 10 cm line with anchor statements ，on the left (no nausea) and on the right (extreme nausea). The patient is asked to mark their current nausea level on the line. The examiner scores the VAS by measuring the distance in either centimeters (0 to 10) or millimeters (0 to 100) from the "no nausea" anchor point.
The first vomiting | 24 hours after surgery
  the time point the first vomiting
The first vomiting's Visual Analogue Scale | 24 hours after surgery
  the Visual Analogue Scale of the first vomiting : the Visual Analog Scale (VAS) is a 10 cm line with anchor statements ，on the left (no vomitting) and on the right (extreme vomiting). The patient is asked to mark their current vomiting level on the line. The examiner scores the VAS by measuring the distance in either centimeters (0 to 10) or millimeters (0 to 100) from the "no vomiting" anchor point.
Total nausea frenquency in postoperative 24 hours | 24 hours after surgery
  the total nausea times of the subjects
The Visual Analogue Scale of nausea in postoperative 24 hours | 24 hours after surgery
  the Visual Analogue Scale of nausea in postoperative 24 hours : the Visual Analog Scale (VAS) is a 10 cm line with anchor statements ，on the left (no nausea) and on the right (extreme nausea). The patient is asked to mark their current nausea level on the line. The examiner scores the VAS by measuring the distance in either centimeters (0 to 10) or millimeters (0 to 100) from the "no nausea" anchor point.
Total vomiting frenquency in postoperative 24 hours | 24 hours after surgery
  the total vomiting times of the subjects
The Visual Analogue Scale of vomiting in postoperative 24 hours | 24 hours after surgery
  the Visual Analogue Scale of vomiting in postoperative 24 hours : the Visual Analog Scale (VAS) is a 10 cm line with anchor statements ，on the left (no vomitting) and on the right (extreme vomiting). The patient is asked to mark their current vomiting level on the line. The examiner scores the VAS by measuring the distance in either centimeters (0 to 10) or millimeters (0 to 100) from the "no vomiting" anchor point.
40-itemquality of recovery score | 24 hours after surgery
  The quality of postoperative life recovery was assessed by questionnaire. The content mainly included five aspects, physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items) and pain (7 items).
Postoperative PONV complications | 30 days after surgery
  The incidence of dizziness, headache, electrolyte imbalance, aspiration, aspiration pneumonia, and wound dehiscence
Postoperative hospital stay | 30 days after surgery
  The interval between the date of discharge and the date of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, MD,PHD, Study Chair — First Affiliated Hospital of Xian JiaotongUniversity
Locations (1):
- First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Gao W, Zhang L, Han X, Wei L, Fang J, Zhang X, Zhang J, Wang H, Zhou Q, Wang C, Chen W, Ni X, Yang L, Du R, Wang G, Liu B, Li Y, Zhang S, Wang Q. Transcutaneous Electrical Acupoint Stimulation Decreases the Incidence of Postoperative Nausea and Vomiting After Laparoscopic Non-gastrointestinal Surgery: A Multi-Center Randomized Controlled Trial. Front Med (Lausanne). 2022 Mar 14;9:766244. doi: 10.3389/fmed.2022.766244. eCollection 2022. PMID 35360742